CLINICAL TRIAL: NCT04875221
Title: Mechanisms of Network-based Real-time fMRI Neurofeedback in Patients With Posttraumatic Stress Disorder
Brief Title: Network-based Neurofeedback in PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study is no longer being conducted by Dr. Lanius - the principal investigator has been changed from Dr. Ruth Lanius to Dr. Andrew Nicholson.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ruth Lanius, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9004
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: PTSD; Post-traumatic Stress Disorder
Keywords: Neurofeedback; NFB
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the experimental or sham arms.
Who Masked: Participant, Investigator
Masking Description: Participants will be randomly assigned to either the experimental or sham-control arms under double-blind conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental neurofeedback arm (Experimental): The experimental arm will be able to view a feedback display that informs them of the strength of connectivity between the target regions. In both arms, feedback signals will be relayed back to the participant in the scanner through visualization software as a thermometer that increases or decreases as the extent to which the neural target model dominates (in other words, as the strength of directed connectivity between regions increases).
  Interventions: Combination Product: Connectivity-based neurofeedback
- Sham-control neurofeedback arm (Sham Comparator): Participants in the sham-control arm will receive yoked sham neurofeedback signal (or fake signal), corresponding to a replayed feedback signal from a successful participant in the experimental group in order to ensure similar motivational states and following standard methods.
  Interventions: Combination Product: Connectivity-based neurofeedback

INTERVENTIONS:
Combination Product: Connectivity-based neurofeedback — Real-time fMRI neurofeedback will be used to non-invasively regulate neural network connectivity patterns associated with symptoms and emotional arousal among patients with PTSD and healthy individuals, with the aim to induce lasting neuronal effects and reduce symptoms.

SUMMARY:
This project will examine the use of real-time fMRI (rt-fMRI) neurofeedback in the regulation of neural networks underlying symptoms experienced by individuals with posttraumatic stress disorder (PTSD). Investigators will use rt-fMRI neurofeedback in order to facilitate emotion regulation during symptom induction, and examine individual differences that influence regulation capacities.

DETAILED DESCRIPTION:
The purpose of this study is to examine the mechanisms of real-time fMRI (rt-fMRI) neurofeedback as a method by which to regulate functional brain connections underlying symptoms/emotions experienced by individuals with PTSD. The aim of this study is to evaluate further the suitability of state-of-the-art fMRI as a non-invasive therapeutic tool among individuals burdened by PTSD, in order to inform future clinical trials of neurofeedback aiming to reduce symptoms of PTSD. This will be achieved by using rt-fMRI and neurofeedback of brain signals, in order to teach individuals with PTSD to self-regulate the neural networks that are associated with their symptoms. Investigators will examine the mechanisms of self-regulating neural networks using real-time neuroimaging and feedback to these brain signals. Neurofeedback is a form of brain training that allows individuals to improve their health by learning to control signals from their own body.

This study will employ a 2 (PTSD group vs. healthy control group) by 2 (arm; experimental vs. sham-control) design. This study involves an assessment which will include clinical interviews and a fMRI (functional magnetic resonance imaging) scan. The fMRI scan will involve trauma-word exposure during neurofeedback task runs. During the presentation of the words in the fMRI scanner, participants in the experimental arm will be able to view a feedback display that informs them of the strength of connectivity between the target regions. Participants in the sham-control arm will receive yoked sham neurofeedback signal (or fake signal), corresponding to a replayed feedback signal from a successful participant in the experimental group in order to ensure similar motivational states and following standard methods. In both arms, feedback signals will be relayed back to the participant in the scanner through visualization software as a thermometer that increases or decreases as the extent to which the target model dominates.

ELIGIBILITY:
Inclusion Criteria:

PTSD Group:

* English speaking
* age: 18-65
* meets diagnostic criteria for PTSD (as determined by study assessment)

Control Group:

* English speaking
* age: 18-65

Exclusion Criteria:

All participants:

* Individuals with any implants, conditions, etc. that do not comply with 3-Tesla fMRI research safety standards (e.g., certain implants, pregnancy)
* history of neurological disorder
* history of any pervasive developmental disorder
* history of significant head injury/lengthy loss of consciousness (e.g., a Glasgow Coma Scale Score < 15 at the time of incident assessed retrospectively by participant)
* significant untreated medical illness
* alcohol/substance abuse or dependence within the last 3 months

PTSD Group:

* history of bipolar disorder
* history of psychosis
* extensive current use of narcotic medications

Control Group:

* any current or past mental health disorders
* extensive current or past psychotherapy
* extensive current or past use of psychotropic or narcotic medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Changes in functional magnetic resonance imaging (fMRI) neural connectivity/activation | 1hour
  Investigators will evaluate changes in fMRI neural connectivity and activation as a function of neurofeedback treatment. Specifically, investigators will evaluate changes in fMRI neural connectivity/activity among brain areas included in the neurofeedback target network (which includes areas within the default mode, salience, and central executive networks).
Changes in emotional experience over neurofeedback training (RSDI scale) | 1-week
  The Response to Script Driven Imagery (RSDI) Scale will assess changes in symptoms after each neurofeedback run in the scanner (3 training runs), in line with previous neurofeedback studies. Investigators will evaluate changes in emotional experience during neurofeedback treatment and at 1-week follow-up, using the RSDI scale. The RSDI has a minimum value of 0 and maximum value of 66 (higher scores indicate more severe symptoms/emotional distress).

SECONDARY OUTCOMES:
Changes in PTSD symptoms over neurofeedback training (PCL-5) | 1-week
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses symptoms of PTSD. The PCL-5 has a variety of purposes, including monitoring symptom change during and after treatment.
  Investigators will evaluate changes in PTSD symptoms from baseline, to post-neurofeedback training and at 1-week follow-up using the PCL-5. The minimum score is 0, the maximum is 80 (higher scores indicate increased PTSD severity).

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A Lanius, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre - University Hospital, London, Onatrio, Canada

IPD SHARING:
Plan to Share IPD: No